CLINICAL TRIAL: NCT00062023
Title: Phase II Study Of Colorectal ACF Screening, Regression And Prevention In High Risk Participants
Brief Title: Comparison of Sulindac, Aspirin, and Ursodiol in Preventing Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed by the NCI.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ID01-454; P30CA016672 (NIH); MDA-ID-01454 (Other: UT MD Anderson Cancer Center); CDR0000304433 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Aspirin; Sulindac; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I Sulindac (Active Comparator): Oral sulindac twice daily.
  Interventions: Drug: Sulindac
- Arm II Aspirin (Active Comparator): Oral aspirin once daily.
  Interventions: Drug: Acetylsalicylic acid (Aspirin)
- Arm III Ursodiol (Active Comparator): Oral ursodiol three times daily.
  Interventions: Drug: Ursodiol
- Arm IV: Sulindac Placebo (Placebo Comparator): Oral sulindac placebo twice daily.
  Interventions: Other: Sulindac Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin) — Patients receive oral aspirin once daily for 12 months.
  Other Names: Aspirin; USAN; ASA
  Arms: Arm II Aspirin
Drug: Sulindac — Patients receive oral sulindac twice daily for 12 months.
  Other Names: Clinoril
  Arms: Arm I Sulindac
Drug: Ursodiol — Patients receive oral ursodiol three times daily for 12 months.
  Other Names: ursodeoxycholic acid; UDCA
  Arms: Arm III Ursodiol
Other: Sulindac Placebo — Oral sulindac placebo twice daily.
  Arms: Arm IV: Sulindac Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. It is not yet known whether sulindac, aspirin, or ursodiol is more effective in preventing colorectal cancer.

PURPOSE: This randomized phase II trial is studying how well sulindac works compared to aspirin or ursodiol in preventing colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the percentage change in colorectal aberrant crypt foci (ACF) in patients with a history of colorectal cancer or at high risk for colorectal cancer when treated with sulindac vs aspirin vs ursodiol.
* Determine the safety and efficacy of these drugs, in terms of ability to cause regression of existing colorectal ACF and prevent new ACF development, in these patients.

OUTLINE: This is a partially blinded, randomized, placebo-controlled study. Patients are stratified according to colorectal neoplasia (adenoma vs carcinoma). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral sulindac twice daily.
* Arm II: Patients receive oral aspirin once daily.
* Arm III: Patients receive oral ursodiol three times daily.
* Arm IV: Patients receive oral sulindac placebo twice daily. In all arms, treatment continues for 12 months in the absence of disease progression or unacceptable toxicity.

Patients undergo a colonoscopy at baseline and at the end of treatment.

Patients are followed at 2 months after the end of treatment.

PROJECTED ACCRUAL: A total of 172 patients (43 per treatment arm) with a history of colorectal cancer or adenomas will be accrued for this study. A total of 20 additional patients with no elevated risk of colorectal neoplasia will be accrued, but not randomized, for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 40-80 years
2. with >5 colorectal ACF and a prior history of colorectal cancer defined as Dukes A/B1 carcinoma within 5 years of entry or any stage of colorectal cancer if at least 5 years post surgical resection (86 subjects)
3. with >5 colorectal ACF and recent/current history of colorectal adenoma(s) defined as one of the following: one adenomatous polyp >1cm or two or more adenomatous polyps of any size or one adenomatous polyp of any size and a documented history of adenomatous polyp(s) (86 subjects)
4. No elevated risk of colorectal cancer or adenomas (20 subjects)
5. Subjects will be permitted to use Nasonex but all other nasal steroids are prohibited. Subjects may change to Nasonex but must have discontinued previous nasal steroid use for at least 30 days prior to study randomization.
6. If participant is female and of childbearing potential, she must agree to use adequate contraception and must have a negative serum pregnancy test within 14 days prior to study drug administration
7. No use of investigational agent(s) within the last 3 months or at the discretion of the medical monitor
8. The subject will be allowed to proceed to randomization so long as all of the following laboratory criteria are met on baseline evaluation: Hgb > 10.0 g/dl, platelet count > 100,000/ul; WBC > 3,000/ul; ALT < 2 x upper limit of normal; AST < 2 x upper limit of normal, and total bilirubin <1.5mg/100ml.
9. Patients requiring use of hormone modulators such as Tamoxifen or Arimidex will be permitted to enroll providing they meet all of the eligibility criteria noted above

Exclusion Criteria:

1. Known diagnosis of FAP, hereditary non-polyposis colon cancer (HNPCC), or inflammatory bowel disease
2. History of hypersensitivity to COX-2 inhibitors, sulfonamides, NSAIDs , salicylates, or ursodeoxycholic acid
3. Use of NSAIDs, including aspirin, at any dose during the six months prior to study entry will require a three month washout period prior to eligibility beginning with the time of the last dose. Participants must be off all NSAIDs for three months prior to study entry. Individuals on cardioprotectant aspirin at any dose will not be eligible.
4. History of gastroduodenal ulcers documented endoscopically would preclude a patient from participation in the trial
5. Known inability to participate in the scheduled follow-up tests.
6. Significant medical or psychiatric problems which would make the patient a poor protocol candidate, in the opinion of the principal investigator.
7. "Unacceptable clinical risk" to proceed (based upon the subclinical discoveries made via baseline colonoscopy and biopsies).
8. Patient has undergone a total colectomy
9. Patient has received chemotherapy within the past 6 months of randomization into study. Topical chemotherapy will be assessed on a case-by-case basis. Any history of pelvic or rectal radiation therapy will exclude a patient from participating.
10. History of invasive carcinoma in the past five years (except patients with Dukes A/B1 carcinoma within 5 years of entry or any stage of colorectal cancer if at least 5 years post surgical resection)
11. Patients with rectal cancer are excluded except for transanal excision without radiation.
12. Patients with acute liver disease, unexplained transaminase elevations or a history of renal stones would be excluded.
13. Participants will not be permitted to be randomized into the trial if any of the following laboratory values are reported at baseline : Hgb < 10.0 g/dl, platelet count <100,000/ul; WBC < 3,000/ul; ALT > 2 x upper limit of normal; AST > 2 x upper limit of normal, and total bilirubin >1.5mg/100ml.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-06; Primary Completion 2005-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Percentage Change in Colorectal ACF Patients Treated with Sulindac, Aspirin or Ursodiol | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Bresalier, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org